CLINICAL TRIAL: NCT05364320
Title: Lumbar Spine Range of Motion and EMG Outcomes in Older Adults
Brief Title: A Study to Evaluate Spine Motion in Older Adults
Acronym: SADLROM
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kenton R. Kaufman, PhD, PE, Principal Investigator, Mayo Clinic
Other Study IDs: 20-013160; K25AG068368 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-05-06 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Men aged 50-64
- Men aged 65 and over
- Women aged 50-64
- Women aged 65 and over

SUMMARY:
This study is being done to measure real-world motions and forces in the spine during everyday activities. This information will be used to develop and validate a computer model of how the spine moves and determine injury risk.

DETAILED DESCRIPTION:
Kinematic motion data will be collected at 120 Hz using a 14-camera Real Time Motion Analysis system. Cortex software (Motion Analysis Corp., Rohnert Park, CA) will be used to visualize the data during physical activities. A developed Matlab code will be used for data analysis. Statistical parametric mapping (SPM) will be used to collect the entire kinematic motion waveforms to compare motion profiles of different individuals. Also, the peak values for each activity will be captured for statistical analysis. Muscle response and electrical activity, which will be used to estimate muscle forces, will be recorded during gait analysis from the paraspinal lumbar muscles using an EMG system. Surface electrodes will be attached to the lumbar spine. EMG data will be collected at 2400 Hz. For each participant, the investigators will record five trials per activity.

Additionally, gait speed as well as static and dynamic balance will assess. Knee and grip strength will also be measured. Finally, physical activity levels will be assessed both objectively and subjectively.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and over
* Ability to perform trunk flexion, lateral bending, and axial rotation, as well as lift at least 5 pounds of weight from the floor

Exclusion Criteria:

* Spinal pathologies
* Physiological and neuromuscular disorders
* BMI>35
* Knee or hip replacement in the past 12 months
* Use of assistive devices
* Frailty: with FRAIL score of 3 or greater

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic's elderly adult patients or residents of Rochester MN with minimum age of 50 years.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Thoracic and lumbar spine ranges of motions in degrees | Day 1
Paraspinal muscle activities in Newtons | Day 1

SECONDARY OUTCOMES:
Upper extremity strength in Newtons | Day 1
Lower extremity strength in Newton-meters | Day 1
Physical activity levels measured by IPAQ questionnaire in MET-minutes per week | Day 1
  MET (metabolic equivalent task) is defined as 1 kcal/kg/hour
Physical activity levels measured by accelerometry in MET-minutes per week | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Kenton Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be stored in the Motion Analysis Lab at Mayo Clinic Rochester.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials